## Statistical analysis

## Statistical analysis

To assess if adding DBT skills to standard treatment is relevant, feasible, accepted and potential

benefits descriptive statistics will be provided. Descriptive statistics for demographic and psychological factors measured on a continuous scale will be reported in terms of mean or median value with appropriate measure on spread (standard deviation or quartiles) whereas the

distribution of categorical factors will be reported in terms of proportions and percentages.